CLINICAL TRIAL: NCT01115023
Title: Randomized Controlled Trial to Study the Effect of Consuming Food Cooked in Iron Utensils on Iron Status in Children With Iron Deficiency Anemia (IDA)
Brief Title: Effect of Consuming Food Cooked in Iron Utensils on Iron Status in Children With Iron Deficiency Anemia (IDA)
Acronym: IDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dhande, Leena Ajay, M.D. (Other)
Collaborators: Sir Gangadharrao Chitnavis Memorial Medical Research Trust Nagpur (Unknown)
Responsible Party: Leena Ajay Dhande, Indira Gandhi Govt Medical College, Nagpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L1IDA1
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2010-04

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia; dietary intervention; To evaluate a cheap and sustainable dietary intervention to improve the iron status of the entire family of the index case of non-severe iron deficiency anemia.
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron group (Experimental): This group received an iron cooking pot for daily household cooking as an intervention
  Interventions: Other: iron cooking pot
- Aluminium group (No Intervention): the subjects in this group were asked to continue cooking in the aluminium pot and not to cook in the iron pot if they possessed one.

INTERVENTIONS:
Other: iron cooking pot — the mother was instructed to cook the family food in the iron cooking pot for the study period (60 days) as frequently in the day as possible.
  Arms: iron group

SUMMARY:
Iron deficiency is a common problem in the world and more so in the developing countries with a prevalence of 64 % (using WHO cut-off values of Hb <11.0 g/dl) among children, 9-36 months of age. The Pediatric population is especially vulnerable to iron deficiency anemia due to low intake of iron rich foods, rapid growth with high demand and losses of iron from body especially with the commonly found worm infestations in children. Mild to moderate iron deficiency is widely prevalent in children and can have several implications including failure to thrive, poor scholastic performance, repeated infections etc. Dietary measures along with therapeutic measures are recommended to combat Iron Deficiency Anemia (IDA). However, iron rich foods alone cannot be relied upon as a sole step to counter IDA. The utensil in which the food is cooked plays a major role in determining the final iron content of food. Several studies have documented that most of the foods (90%) contained significantly more iron when cooked in iron utensils depending on the acidity, moisture content, and cooking time of food.The daily dietary intake could vary from 11 to 6 mg of iron if iron utensil was used for cooking [3].

Food cooked in Aluminum (Al) utensils has a higher Al content which can be detrimental to healthy individuals and particularly to patients with chronic renal failure.In healthy persons, diseases of central nervous system, as well as of hematopoeitic system, skeletal system and respiratory system are described due to excess of Aluminium consumption. Aluminium utensils have fast replaced iron cooking pots from Indian kitchens, hence a study to know the effectiveness of iron cooking pot as a measure to combat IDA is necessary.

Studies have shown the utility of cooking food in iron utensil in prevention of IDA but the investigators did not come across a study to document the use of this modality in treatment of IDA in children. Since the investigators anticipate that the improvement of iron status will be a gradual process, so the investigators decided to evaluate the utility of cooking food in iron utensils on iron status in children with non-severe IDA (Hb% < cutoff point for age but > 5 gm %.

To test the following hypothesis "use of iron utensils for cooking food will result in improvement in iron status in Pediatric patients with nonsevere Iron Deficiency Anemia."

DETAILED DESCRIPTION:
Dietary advice and iron therapy are considered the cornerstones of treating a patient with non-severe IDA. The foods that are rich in Iron include meat and poultry products, egg, green leafy vegetables, jaggery, dry fruits etc. Iron in food is of two types viz. haem iron and non haem iron. Haem Iron has excellent bioavailability but the bioavailability of the non-haem Iron in the food stuffs is considerably affected by the presence of substances like phosphates, phytates, tannins and fibres. On the other hand, Ascorbic acid, sugars and other acidic substances in the food enhance the iron absorption. The bulk of food consumed by a child is too less to provide him with therapeutic amounts of iron form diet alone. In the developing countries, the child is quite unlikely to get poultry products and meat as a source of haem Iron. If in this situation, the child is provided with food cooked in Iron utensil, then it provides additional Iron to meet the increased demand. This will not only be cost effective but it will also alter the cooking practices and thereby have a long term effect on the iron status of the entire family. Thus it will treat the IDA in the index case and will also benefit other family members who may be having borderline or overt iron deficiency. This cost effective measure if incorporated in the health policy of the country will certainly have widespread positive implications on the health of the general population.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria

1. Age: 2-12 years,
2. Resident of urban Nagpur
3. Diagnosed as having non-severe IDA defined as Hb% > 5gm% but less than cut off point for age for diagnosing anemia.

Exclusion Criteria:

1. Suffering from Hemoglobinopathy or Iron overload due to any cause
2. Receiving Iron therapy
3. Malabsorption
4. Bleeding diathesis
5. Chronic illness
6. Participation in another trial in last 30 days

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2003-10; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
to compare the rise in Hemoglobin at the end of 60 days period in the iron group vs the aluminium group. | 60 days

SECONDARY OUTCOMES:
to compare the change in RDW, RBC indices and Reticulocyte count at the end of 60 days period in the iron group vs the aluminium group. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Leena Ajay Dhande, MD (Pediatrics), Principal Investigator — Associate Professor
Locations (1):
- Government Medical College, Nagpur, Maharashtra, India